CLINICAL TRIAL: NCT02387788
Title: Phase 2a Open Label Study to Assess the Efficacy and Safety of Subcutaneous 15mg AKB-9778 Administered Twice Daily for 84 Days in Subjects With Retinal Vein Occlusion
Brief Title: Open Label Study to Assess the Efficacy and Safety of AKB-9778 in Subjects With Macular Edema Due to RVO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerpio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKB-9778-CI-4001
Record Dates: First submitted 2015-03-05; First posted 2015-03-13 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — AKB-9778

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 15 mg AKB-9778 BID for 84 days (Experimental): Subcutaneous AKB-9778 15 mg BID (total dose of 30 mg/day) for 84 days
  Interventions: Drug: AKB-9778

INTERVENTIONS:
Drug: AKB-9778 — Phase 2a open-label study to assess the efficacy and safety of subcutaneous 15mg AKB-9778 administered twice daily for 84 days in subjects with macular edema due to RVO.

SUMMARY:
Phase 2a open-label study to assess the efficacy and safety of subcutaneous 15mg AKB-9778 administered twice daily for 84 days in subjects with macular edema due to RVO.

DETAILED DESCRIPTION:
Subjects will participate in the study for up to 168 days. Up to 20 subjects will be enrolled in the study.

Subjects will self-administer study medication as subcutaneous (SC) injections in the abdomen (preferably) twice per day; the first dose each day should be administered in the morning and the evening dose should be administered within 8 to 16 hours after the morning dose.

Safety assessments will be conducted at each study visit during treatment and AEs will be collected throughout the Treatment period and during the 56-days observation period visits.

ELIGIBILITY:
The following is a abbreviated list of Inclusion Criteria:

* Definite retinal thickening due to RVO involving the central macula based on Investigator's clinical evaluation and demonstrated by sdOCT.
* Mean central subfield thickness of at least 300 µm by sdOCT with presence of intraretinal fluid
* ETDRS BCVA letter score ≤ 76 and ≥ 24.
* Decrease in vision determined to be primarily the result of macular dema due to RVO and not due to other causes.

The following is a abbreviated list of Exclusion Criteria:

* Macular edema is considered to be due to a cause other than RVO
* Any other ocular disease that may cause substantial reduction in visual acuity, including iris neovascularization, retinal detachment, epiretinal membrane, vitreous hemorrhage or fibrosis, ocular inflammation (uveitis), retinal inflammatory, infectious disease, or primary open-angle glaucoma.
* High myopia (-8 diopter or more correction).
* History of idiopathic or autoimmune uveitis.
* History of any ocular surgery within 3 months prior to Day 1.
* History of panretinal scatter photocoagulation (PRP) or focal laser within 3 months prior to Day 1.
* History of prior intravitreal, subtenon, or periocular steroid therapy within 3 months prior to Day 1 (e.g., triamcinolone).
* History of prior treatment with intravitreal anti-VEGF treatment within 16 weeks prior to Day 1.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Visual acuity in subjects with RVO | 84 days
  Best corrected visual acuity is measured by ETDRS charts

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Campochiaro, MD, Principal Investigator — Wilmer Eye Institute
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No